CLINICAL TRIAL: NCT03074994
Title: The Comparative Efficacy of Peri-articular and Intraarticular Tranexamic Acid in Total Knee Arthroplasty: A Prospective, Double-Blind Randomized, Controlled Trial
Brief Title: The Comparative Efficacy of Peri-articular and Intraarticular Tranexamic Acid in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thammasat University (Other)
Collaborators: Boontanapibul, Krit, M.D. (Individual)
Responsible Party: Principal Investigator, piya pinsornsak, Principal Investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MTU-EC-OT-6-063/59
Record Dates: First submitted 2016-11-20; First posted 2017-03-09 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2018-06

CONDITIONS: Osteoarthritis,Knee
Keywords: Tranexamic acid; Peri-articular injection; Intraarticular injection; Total knee arthroplasty; Blood loss
MeSH Terms: conditions — Osteoarthritis, Knee; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Peri-articular tranexamic acid injection (Experimental): TXA combined with multimodal local anesthetic infiltration inject into peri-articular area (Anterior soft tissue+Medial gutter area+Lateral gutter area)
  Interventions: Drug: Peri-articular TXA (15 mg/kg); Procedure: TXA combined with multimodal local anesthetic infiltration inject into peri-articular area
- Intraarticular tranexamic acid injection (Experimental): TXA inject into intraaricular knee capsule after multimodal local anesthetic infiltration
  Interventions: Drug: Intraarticular TXA 2 g (40 mL); Procedure: TXA 40 mL inject into intraaricular knee capsule
- Control group (No Intervention): Don't receive any route of TXA

INTERVENTIONS:
Drug: Peri-articular TXA (15 mg/kg) — combined with multimodal local anesthetic infiltration (0.5% bupivacaine 100 mg, morphine sulfate 5 mg, 0.1% epinephrine 0.6 mg, and ketorolac 30 mg) mixed NSS up to 75 mL
  Arms: Peri-articular tranexamic acid injection
Drug: Intraarticular TXA 2 g (40 mL) — inject separate from multimodal local anesthetic infiltration (0.5% bupivacaine 100 mg, morphine sulfate 5 mg, 0.1% epinephrine 0.6 mg, and ketorolac 30 mg mixed NSS up to 75 mL)
  Arms: Intraarticular tranexamic acid injection
Procedure: TXA combined with multimodal local anesthetic infiltration inject into peri-articular area — (Anterior soft tissue 25 mL+Medial gutter area 25 mL+Lateral gutter area 25 mL) prior to capsular closure and tourniquet deflation
  Arms: Peri-articular tranexamic acid injection
Procedure: TXA 40 mL inject into intraaricular knee capsule — after multimodal local anesthetic infiltration (Anterior soft tissue 25 mL+Medial gutter area 25 mL+Lateral gutter area 25 mL) prior to tourniquet deflation
  Arms: Intraarticular tranexamic acid injection

SUMMARY:
Post-operative bleeding in total knee arthroplasty (TKA) can result in hypovolemic shock and unnecessity for allogenic blood transfusions. Intravenous and topical tranexamic acid (TXA) have been well established in reducing blood loss postoperatively. However, there are lack of data on peri-articular TXA injection during TKA. Therefore, the investigators conducted a three-arm prospective, randomized, controlled trial to compare the effectiveness of bleeding reduction of peri-articular TXA injections, intraarticular TXA injections and control group.

DETAILED DESCRIPTION:
Patients scheduled for unilateral primary TKA; 108 patients were randomly assigned to receive peri-articular TXA, intraarticular TXA and control group. 36 patients received either: (I) 15 mg/kg peri-articular TXA combined with multimodal local anesthetic infiltration (bupivacaine, morphine, ketorolac and epinephrine) into the anterior soft tissue, medial gutter area, lateral gutter area prior to capsular closure and tourniquet deflation (group 1). (II) 2 g of intraarticular TXA after complete capsular closure just before tourniquet deflation (group 2). (III) Don't receive any route of TXA in control group (group 3). Hemoglobin (Hb) concentrations were measured at 24 and 48 hour, and the number of blood transfusions and knee circumference measurements were recorded. Serum TXA was recorded at 2 and 24 hours after operation. The reviewers were blinded to treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with osteoarthritis in need of a TKA

Exclusion Criteria:

* Inflammatory arthritis
* Post-traumatic arthritis
* A history of or current venous thromboembolic disease
* Any underlying disease of haemostasis, cirrhosis, chronic renal failure, patients on anticoagulants or strong antiplatelet drugs (e.g. warfarin, clopidogrel)
* Preoperative hemoglobin <10 g/dL or a platelet count < 140,000 /uL3
* Allergy to TXA

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline hemoglobin concentrations | 48 hours after the operation
Unit of blood transfusion | 48 hours after the operation

SECONDARY OUTCOMES:
Tranexamic acid level in blood | 2 and 24 hours after the operation
Knee diameter for swelling | 24 and 48 hours after the operation
Local soft tissue complications | 14 days after the operation
Skin necrosis | 24 and 48 hours after the operation
Number of patient with venous thromboembolism | 14 days after the operation
Visual Analogue Scales | 24 and 48 hours after the operation
  (VAS, 0 = no pain, 10 = the worst imaginable pain)
Knee flexion angle | 24 and 48 hours after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat university hospital, Pathum Thani, Klongluang, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Madjdpour C, Spahn DR. Allogeneic red blood cell transfusions: efficacy, risks, alternatives and indications. Br J Anaesth. 2005 Jul;95(1):33-42. doi: 10.1093/bja/aeh290. Epub 2004 Oct 14. PMID 15486006
- [Result] Fiebig E. Safety of the blood supply. Clin Orthop Relat Res. 1998 Dec;(357):6-18. doi: 10.1097/00003086-199812000-00003. PMID 9917695
- [Result] Heddle NM, Klama LN, Griffith L, Roberts R, Shukla G, Kelton JG. A prospective study to identify the risk factors associated with acute reactions to platelet and red cell transfusions. Transfusion. 1993 Oct;33(10):794-7. doi: 10.1046/j.1537-2995.1993.331094054613.x. PMID 8236418
- [Result] Juelsgaard P, Larsen UT, Sorensen JV, Madsen F, Soballe K. Hypotensive epidural anesthesia in total knee replacement without tourniquet: reduced blood loss and transfusion. Reg Anesth Pain Med. 2001 Mar-Apr;26(2):105-10. doi: 10.1053/rapm.2001.21094. PMID 11251132
- [Result] Sharma V, Fan J, Jerath A, Pang KS, Bojko B, Pawliszyn J, Karski JM, Yau T, McCluskey S, Wasowicz M. Pharmacokinetics of tranexamic acid in patients undergoing cardiac surgery with use of cardiopulmonary bypass. Anaesthesia. 2012 Nov;67(11):1242-50. doi: 10.1111/j.1365-2044.2012.07266.x. Epub 2012 Jul 24. PMID 22827564
- [Result] Alshryda S, Sarda P, Sukeik M, Nargol A, Blenkinsopp J, Mason JM. Tranexamic acid in total knee replacement: a systematic review and meta-analysis. J Bone Joint Surg Br. 2011 Dec;93(12):1577-85. doi: 10.1302/0301-620X.93B12.26989. PMID 22161917
- [Result] Yang ZG, Chen WP, Wu LD. Effectiveness and safety of tranexamic acid in reducing blood loss in total knee arthroplasty: a meta-analysis. J Bone Joint Surg Am. 2012 Jul 3;94(13):1153-9. doi: 10.2106/JBJS.K.00873. PMID 22623147
- [Result] Zhang H, Chen J, Chen F, Que W. The effect of tranexamic acid on blood loss and use of blood products in total knee arthroplasty: a meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2012 Sep;20(9):1742-52. doi: 10.1007/s00167-011-1754-z. Epub 2011 Nov 8. PMID 22065294
- [Result] Ho KM, Ismail H. Use of intravenous tranexamic acid to reduce allogeneic blood transfusion in total hip and knee arthroplasty: a meta-analysis. Anaesth Intensive Care. 2003 Oct;31(5):529-37. doi: 10.1177/0310057X0303100507. PMID 14601276
- [Result] Panteli M, Papakostidis C, Dahabreh Z, Giannoudis PV. Topical tranexamic acid in total knee replacement: a systematic review and meta-analysis. Knee. 2013 Oct;20(5):300-9. doi: 10.1016/j.knee.2013.05.014. Epub 2013 Jun 28. PMID 23815893
- [Result] Wang H, Shen B, Zeng Y. Comparison of topical versus intravenous tranexamic acid in primary total knee arthroplasty: a meta-analysis of randomized controlled and prospective cohort trials. Knee. 2014 Dec;21(6):987-93. doi: 10.1016/j.knee.2014.09.010. Epub 2014 Oct 23. PMID 25450009
- [Result] Wong J, Abrishami A, El Beheiry H, Mahomed NN, Roderick Davey J, Gandhi R, Syed KA, Muhammad Ovais Hasan S, De Silva Y, Chung F. Topical application of tranexamic acid reduces postoperative blood loss in total knee arthroplasty: a randomized, controlled trial. J Bone Joint Surg Am. 2010 Nov 3;92(15):2503-13. doi: 10.2106/JBJS.I.01518. PMID 21048170
- [Result] Jain NP, Nisthane PP, Shah NA. Combined Administration of Systemic and Topical Tranexamic Acid for Total Knee Arthroplasty: Can It Be a Better Regimen and Yet Safe? A Randomized Controlled Trial. J Arthroplasty. 2016 Feb;31(2):542-7. doi: 10.1016/j.arth.2015.09.029. Epub 2015 Sep 26. PMID 26507526
- [Result] Konig G, Hamlin BR, Waters JH. Topical tranexamic acid reduces blood loss and transfusion rates in total hip and total knee arthroplasty. J Arthroplasty. 2013 Oct;28(9):1473-6. doi: 10.1016/j.arth.2013.06.011. Epub 2013 Jul 23. PMID 23886406
- [Result] Ker K, Beecher D, Roberts I. Topical application of tranexamic acid for the reduction of bleeding. Cochrane Database Syst Rev. 2013 Jul 23;2013(7):CD010562. doi: 10.1002/14651858.CD010562.pub2. PMID 23881695
- [Result] Winter SF, Santaguida C, Wong J, Fehlings MG. Systemic and Topical Use of Tranexamic Acid in Spinal Surgery: A Systematic Review. Global Spine J. 2016 May;6(3):284-95. doi: 10.1055/s-0035-1563609. Epub 2015 Sep 21. PMID 27099820
- [Result] Pinsornsak P, Rojanavijitkul S, Chumchuen S. Peri-articular tranexamic acid injection in total knee arthroplasty: a randomized controlled trial. BMC Musculoskelet Disord. 2016 Jul 26;17:313. doi: 10.1186/s12891-016-1176-7. PMID 27455842
- [Result] Callaghan JJ, O'Rourke MR, Liu SS. Blood management: issues and options. J Arthroplasty. 2005 Jun;20(4 Suppl 2):51-4. doi: 10.1016/j.arth.2005.03.018. PMID 15991130
- [Result] Sa-ngasoongsong P, Chanplakorn P, Wongsak S, Uthadorn K, Panpikoon T, Jittorntam P, Aryurachai K, Angchaisukisiri P, Kawinwonggowit V. An In Vivo Study of Low-Dose Intra-Articular Tranexamic Acid Application with Prolonged Clamping Drain Method in Total Knee Replacement: Clinical Efficacy and Safety. Biomed Res Int. 2015;2015:164206. doi: 10.1155/2015/164206. Epub 2015 Oct 25. PMID 26583092
- [Result] Chang CH, Chang Y, Chen DW, Ueng SW, Lee MS. Topical tranexamic acid reduces blood loss and transfusion rates associated with primary total hip arthroplasty. Clin Orthop Relat Res. 2014 May;472(5):1552-7. doi: 10.1007/s11999-013-3446-0. Epub 2014 Jan 3. PMID 24385043